CLINICAL TRIAL: NCT02316639
Title: The Effectiveness of Neuromuscular Training in Healthy and ACL-Injured Adolescent Females
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Jason Peeler, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H2014:302
Record Dates: First submitted 2014-09-16; First posted 2014-12-15 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: ACL-injury
Keywords: Neuromuscular Training; Skeletally Immature; Knee Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular Training - No Exercise (Experimental): Subjects will participate in 5 weeks of neuromuscular training followed by 5 weeks of no exercise intervention
  Interventions: Other: Neuromuscular Training
- No Exercise - Neuromuscular Training (Experimental): No exercises will be administered for 5 weeks, followed by 5 weeks of neuromuscular Training.
  Interventions: Other: Neuromuscular Training

INTERVENTIONS:
Other: Neuromuscular Training — The established Neuromuscular Training (NMT) protocol is supervised, progressive program in which the patient maintains balance on three different support surfaces while a clinician administers purposeful manipulations of the support system.1 The patient maintains a single-leg stance on the rollerboard and tiltboard surfaces, and a two-leg stance with one foot on a roller board while the other is on a platform. Participants will complete two training sessions per week, for five weeks for a total of 10 training sessions.

SUMMARY:
Recently, there has been a dramatic rise in the number of children participating in competitive sports. Adolescents involved in sports that require cutting, pivoting or body contact are at greatest risk for sustaining an anterior cruciate ligament (ACL) rupture of the knee, however, appropriate management remains controversial. The surgical technique is commonly performed in the adult population has been associated with risks for growth disturbance when performed on skeletally immature individuals. Therefore, the recommended standard of care in children is to initially follow a non-surgical management protocol that allows a patient to skeletally mature prior to ultimately receiving surgical reconstruction. Unfortunately, current non-surgical management protocols are ineffective at enhancing knee joint stability and dynamic function. There has been no research to indicate the most appropriate exercise program for the ACL deficient skeletally immature individual. A neuromuscular exercise program proven to be safe and effective in the ACL deficient adult population is perturbation training. In adolescents, research suggests neuromuscular exercises can reduce the rate of ACL injuries by 50%. However, currently there is no research investigating the benefits of a neuromuscular exercise on the management of a skeletally immature ACL-deficient individual. The results of this investigation will provide researchers and clinicians valuable information on the effect of neuromuscular perturbation exercises on knee joint stability and function immediately following injury. This has the potential to minimize the development of secondary meniscal tears and premature joint degeneration commonly demonstrated following an ACL injury.

DETAILED DESCRIPTION:
Following ethics approval by the University of Manitoba and the Winnipeg Regional Health Authority, 44 participants will be recruited for the study. During the intake session, subjects will complete informed and assent consent, participant information and knee demographic forms. A radiographic report of the knee confirming that the subject is skeletally immature will be obtained from the referring orthopedic surgeon or performed at the Pan Am clinic. For only the ACL-injured subjects, a clinical examination diagnosis and KT-1000 test will confirm the injury. Anthropometric data, such as age, height, weight, range of motion, leg circumference and the pubertal maturation observation scale (PMOS), will be collected. All subjects are required to pass the standardized screening protocol prior to continuing with the testing procedures.

Testing Sessions:

Each subject will participate in 4 follow-up test sessions after the initial intake; Pre-exercise session at the start of the study, Follow-up #1 at the mid-point of the study, Follow-up #2 at the end of the study and a Test-retest session during the no exercise phase of the study. Within the same week as completing the intake session, all subjects will complete the pre-exercise test session. All follow-up testing sessions will include: 1. Subjective evaluation of knee function via the Pedi-IKDC and Physical Activity Questionnaire for Children (PAQ-C), 2. Standardized warm-up on a stationary bike, 3. Dynamic balance evaluation using the SEBT and Y-Balance tests, 4. Strength testing using the Biodex isokinetic dynamometer and core stability tests, and 5. Knee laxity testing using the KT-1000. Both ACL-injured and healthy knee subjects will be randomly divided into two groups, Group A & B. The week following baseline testing, Group A will begin the 5-week NMT protocol, complete a follow-up #1 testing session, then receive no intervention for 5 weeks, and return for a follow-up #2 testing session. The week following baseline testing, Group B will receive of no intervention for 5 weeks, then complete a follow-up #1 test session, complete the 5-week NMT protocol and then return for a follow-up #2 testing session. The test-retest session will be conducted during the first week of the "No Exercise" phase.

Neuromuscular Training (NMT) Sessions:

The established Neuromuscular Training (NMT) protocol is supervised, progressive program in which the patient maintains balance on three different support surfaces while a clinician administers purposeful manipulations of the support system.1 The patient maintains a single-leg stance on the rollerboard and tiltboard surfaces, and a two-leg stance with one foot on a roller board while the other is on a platform. Participants will complete two training sessions per week, for five weeks for a total of 10 training sessions. During each session, both legs will receive training for 2-3 sets of 1 minute duration on each of the support surfaces. Subjects will complete all training sessions with a Certified Athletic Therapist or Physiotherapist at the Pan Am clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 10-14.
2. Radiographic evidence of skeletally immaturity at the knee joint.
3. ACL-injured patients require a clinical examination and a KT-1000 test of > 3mm compared with the contralateral knee to confirm a uni-lateral ACL injury diagnosis.
4. Pass the standardized screening protocol, which includes:

   i. No evidence of joint effusion via swipe test ii. Full passive knee joint range of motion iii. Full active knee extension during a straight leg raise test iv. Quadriceps femoris maximum voluntary isometric contraction force on the involved limb equivalent to 75% of that on the uninvolved limb v. Tolerance for 10 consecutive single-leg hops on the involved limb without pain.

Exclusion Criteria:

1. Symptomatic meniscus or concomitant knee ligament injuries.
2. Recent history (within the 6 months) of a traumatic head (concussion), hip, knee or ankle injury.
3. Reports more than one episode of the knee giving way or buckling resulting in pain and joint effusion from the time of injury. The mechanism at the time of injury is not included.
4. Actively participating in another rehabilitation protocol during the course of the study.
5. Unwillingness or inability to return for follow-up test sessions.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Star Excursion Balance Test (SEBT) at week 7 | week 7
  The SEBT is a valid and reliable non-instrumented test to evaluate dynamic balance in healthy and ACL-injured subjects, however use in the skeletally immature population is lacking in the literature. The subjects perform a series of single-limb squats using the non-stance limb to reach maximally to touch a point along 1 of 8 designated lines on the ground. The reach distance is normalized to the subject's leg length to allow comparison of performance between limbs (injured vs non-injured), between subjects (healthy vs ACL-injured) and before & after an intervention to quantify deficits or improvements in dynamic postural-control. Subjects will perform 4 familiarization trials in each direction, as indicated by previous research. Both limbs will be tested in each direction with the average of the 3 test trails being used for data analysis.

SECONDARY OUTCOMES:
Change from baseline in Y-Balance Test at week 7 | week 7
  The Y-balance test is a commercially available product that evaluates three components of the SEBT. The instrumented version was designed to improve the efficiency of the SEBT. Subjects maintain a one-leg stance on an elevated stance platform from which 3 pieces of plastic pipe extend in the anterior, posteromedial and posterolateral reach directions. With the non-stance foot participants push an indicator to a maximum distance along the pipe, which is marked with 5mm increments. Research indicates that the test is a feasible and reproducible measure of dynamic postural control in children, as well as adults, however testing within the ACL-injured population is lacking. Following the standardized testing procedures, 6 familiarization trials will be performed prior to collecting data for the test trials. The average maximal reach distance for each direction will be used for data analysis.
Change from baseline in Y-Balance Test at week 13 | week13
  The Y-balance test is a commercially available product that evaluates three components of the SEBT. The instrumented version was designed to improve the efficiency of the SEBT. Subjects maintain a one-leg stance on an elevated stance platform from which 3 pieces of plastic pipe extend in the anterior, posteromedial and posterolateral reach directions. With the non-stance foot participants push an indicator to a maximum distance along the pipe, which is marked with 5mm increments. Research indicates that the test is a feasible and reproducible measure of dynamic postural control in children, as well as adults, however testing within the ACL-injured population is lacking. Following the standardized testing procedures, 6 familiarization trials will be performed prior to collecting data for the test trials. The average maximal reach distance for each direction will be used for data analysis.
Change from baseline in Star Excursion Balance Test at week 13 | week 13
  The SEBT is a valid and reliable non-instrumented test to evaluate dynamic balance in healthy and ACL-injured subjects, however use in the skeletally immature population is lacking in the literature. The subjects perform a series of single-limb squats using the non-stance limb to reach maximally to touch a point along 1 of 8 designated lines on the ground. The reach distance is normalized to the subject's leg length to allow comparison of performance between limbs (injured vs non-injured), between subjects (healthy vs ACL-injured) and before & after an intervention to quantify deficits or improvements in dynamic postural-control. Subjects will perform 4 familiarization trials in each direction, as indicated by previous research. Both limbs will be tested in each direction with the average of the 3 test trails being used for data analysis.

OTHER OUTCOMES:
Change from baseline in Quadriceps and Hamstring Strength at week 7 | week 7
  Isometric and Isotonic strength of leg & hip musculature will be assessed with dynamometry.
Change from baseline in Quadriceps and Hamstring Strength at week 13 | week 13
  Isometric and Isotonic strength of leg & hip musculature will be assessed with dynamometry.
Change from baseline in Pedi- International Knee Documentation Committee (IKDC) score at week 7 | week 7
  The pedi-IKDC is a knee-specific measure of symptoms, function and sports activity developed specifically for use in children and adolescents, ages 10-18. The pedi-IKDC has demonstrated acceptable validity, reliability and responsiveness with various knee disorders.
Change from baseline in Pedi-IKDC score at week 13 | week 13
  The pedi-IKDC is a knee-specific measure of symptoms, function and sports activity developed specifically for use in children and adolescents, ages 10-18. The pedi-IKDC has demonstrated acceptable validity, reliability and responsiveness with various knee disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Peeler, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada